CLINICAL TRIAL: NCT00490113
Title: Effects of Pyridoxamine on Oxalate Excretion in Stone Disease and Hyperoxaluria
Brief Title: A Trial of Pyridoxamine to Lower Urine Oxalate in Subjects With Stone Disease or Hyperoxaluria
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Drug unavailable
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 10417; 1R21DK072454-02 (NIH)
Record Dates: First submitted 2007-06-20; First posted 2007-06-22 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Kidney Stones
MeSH Terms: conditions — Kidney Calculi | interventions — Pyridoxamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Pyridoxamine

INTERVENTIONS:
Drug: Pyridoxamine — Two 250 mg capsules, or placebo, given twice a day for four, 4 week periods. Subjects with primary hyperoxaluria will aslo receive escalated doses up to 3500 mg/day for up to 6 1/2 days.

SUMMARY:
To determine whether pyridoxamine can decrease oxalate excretion in subjects who have normal oxalate excretion (but who have had kidney stones), and in subjects who have primary hyperoxaluria.

ELIGIBILITY:
Inclusion Criteria:

* Adults > 18 years
* History of stone formation
* Good Renal function
* Normal urinary excretion of stone-promoting chemicals(Ca, uric acid, oxalate, citrate), except for subjects with hyperoxaluria for Study

Exclusion Criteria:

* Pregnancy
* Hyperparathyroidism
* Enteric hyperoxaluria.
* Obstructive uropathy
* Infection (struvite) stones
* Severe dietary Ca++ restriction or deficiency
* Recent significant cardio-vascular events

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-01

PRIMARY OUTCOMES:
Urinary Excretion of Oxalate at Highest Dose | 4 Weeks

SECONDARY OUTCOMES:
Change in Urinary Supersaturation | 4 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jon I Scheinman, M.D., Principal Investigator — University of Kansas Medical Center